CLINICAL TRIAL: NCT00500526
Title: Effects of Singing on Dyspnea, Quality of Life and Pulmonary Function Parameters of COPD Patients in Stable Conditions.
Brief Title: Effects of Singing in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4626/2004HCFMRP-USP
Record Dates: First submitted 2007-07-11; First posted 2007-07-12 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Pulmonary function; Respiratory muscle; Dyspnea; Quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Singing Group (Experimental): Patients who will receive singing classes
  Interventions: Other: Singing practice; Other: Singing classes
- 2 Control group (Other): Patients who will attend hand craft classes
  Interventions: Other: Hand craft classes

INTERVENTIONS:
Other: Singing practice
  Arms: 1 Singing Group
Other: Singing classes
  Arms: 1 Singing Group
Other: Hand craft classes
  Arms: 2 Control group

SUMMARY:
The purpose of this study is to investigate the effects of the practice of singing for a long period of time on pulmonary function data, quality of life, and dyspnea sensation of patients with COPD in stable clinical conditions. As singing is a type of respiratory training, the study hypothesis is that singing would improve maximal respiratory pressures, dyspnea sensation, and overall quality of life of these patients.

DETAILED DESCRIPTION:
Thirty COPD patients in stable clinical conditions are going to be randomized in two groups: the first one is going to have singing classes for six months; the other one is going to have classes of general manual arts for a similar period of time. The patients of both groups are going to perform spirometry, measurements of maximal respiratory pressures and answer the health related quality of life questionnaires SF-36 and Saint George's before the beginning of practice and after 6 months.Both singing and manual arts practices are going to be administered one hour a week by specialized teachers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD according GOLD criteria
* Stable clinical conditions for the previous two months

Exclusion Criteria:

* Severe comorbidities other than COPD
* Hypoxemia with partial arterial oxygen pressure lower than 50 mmHg
* Incapacity to come to the research center in a weekly basis.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Forced vital capacity, forced expiratory volume, functional residual capacity, inspiratory capacity, maximal respiratory pressures | 6 months

SECONDARY OUTCOMES:
General quality of life score: SF-36 questionnaire.Specific quality of life score : Saint George's Questionnaire; Basal dyspnea index | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: José B Martinez, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clínicas de Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Bonilha AG, Onofre F, Vieira ML, Prado MY, Martinez JA. Effects of singing classes on pulmonary function and quality of life of COPD patients. Int J Chron Obstruct Pulmon Dis. 2009;4:1-8. Epub 2009 Apr 15. PMID 19436683